CLINICAL TRIAL: NCT00198861
Title: Neurobehavioral Model of HIV in Injection Drug Users
Status: Completed | Type: Observational
Sponsor: The City College of New York (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Dr. William Latimer, Professor and Dean, The City College of New York
Other Study IDs: 5R01DA014498-05 (NIH); 5R01DA014498 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-08

CONDITIONS: Drug Abuse; HIV Infections
Keywords: HIV Epidemiology; Neurology; Neuropsychological; HIV Risk Factors; Cognitive Risk Factors; HIV
MeSH Terms: conditions — Substance-Related Disorders; HIV Infections | interventions — Injections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Injection and Non-Injection Drug Users: (1) the degree to which specific executive dysfunctions predispose heroin and cocaine users to high-risk injection practices or sex behaviors, and (2) whether observed relationship between executive dysfunction and HIV-risk behaviors can be understood independent of levels of drug -taking frequency, or whether the observed data are more consistent with complex patterns of interdependency between executive dysfunction, drug-taking frequency, and HIV-risk-behaviors
  Interventions: Other: Injection and Non-Injection Drug Users

INTERVENTIONS:
Other: Injection and Non-Injection Drug Users — (1) the degree to which specific executive dysfunctions predispose heroin and cocaine users to high-risk injection practices or sex behaviors, and (2) whether observed relationship between executive dysfunction and HIV-risk behaviors can be understood independent of levels of drug -taking frequency, or whether the observed data are more consistent with complex patterns of interdependency between executive dysfunction, drug-taking frequency, and HIV-risk-behaviors.

SUMMARY:
The purpose of this R01 study is to evaluate the association between neuropsychological executive dysfunction and HIV infection among young injection and non-injection drug users. A longitudinal study will be conducted in which the cohort of seronegative drug users completing a baseline neuropsychological battery are re-assessed on three subsequent occasions, roughly six months apart. The primary aim of the longitudinal study is to estimate the magnitude of the suspected causal relationship between executive dysfunction and HIV-risk behaviors while adjusting for time-invariant (e.g. sex, ethnicity) and time-varying (e.g. degree of drug abuse) covariates. We also seek to evaluate: (1) the degree to which specific executive dysfunctions predispose heroin and cocaine users to high-risk injection practices or sex behaviors, and (2) whether observed relationship between executive dysfunction and HIV-risk behaviors can be understood independent of levels of drug -taking frequency, or whether the observed data are more consistent with complex patterns of interdependency between executive dysfunction, drug-taking frequency, and HIV-risk-behaviors. If successful, this project will shed new light on significant and potentially malleable HIV-risk factors in injection and non-injection drug users. This will be important evidence because injection drug abuse continues to account for a large proportion of HIV seroconversions particularly among young women and minorities. As such, this RO1 research project serves as an important initial step in a line of innovative investigations about suspected causal associations between neuropsychological deficits and HIV-risk behaviors in drug users. Ultimately, this line of investigation should lead to changes in public and clinical practices designed to prevent HIV infection.

ELIGIBILITY:
Inclusion Criteria:

* Drug users aged 15 to 50 years old.

Exclusion Criteria:

* Acute psychotic, suicidal, homicidal ideation.

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: In total, we seek to recruit 150 HIV positive and 800 HIV negative drug users who are between the ages of 15 and 50 years and who have used illicit drugs within the previous five years of enrollment.
Sampling Method: Probability Sample
Enrollment: 836 (Actual)
Dates: Start 2002-02; Primary Completion 2015-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
HIV-Risk Behavior Outcomes | Outcome measure will be assessed at 6, 12 , and up to 18 months after enrollment.
  Among the drug-related HIV-risk behaviors are drug use cessation and relapse, risky injection practices, including direct and indirect syringe sharing, disinfection practices, and injection in high risk contexts (e.g. shooting galleries). Sexual practices include number and types of partners (gender), type(s) of sexual acts (oral, vaginal and anal intercourse), condom use, survival sex (sex for money, drugs, shelter, food and protection), and incident sexually transmitted diseases.

SECONDARY OUTCOMES:
Executive Functions | Outcome measure will be assessed at 6, 12 , and up to 18 months after enrollment.
  Executive function measures will be derived for working memory, response inhibition, planning, decision making, and conceptual reasoning/cognitive flexibility. A measure of working memory may be derived from the Digits Backward portion of the WAIS-III Digit Span subtest. Components of response inhibition will be assessed by a Go No-Go task that measures impulse control and the Stroop Color-Word Test that measures interference control. A measure of impulse control may be derived from the errors of commission score from the Go No-Go task.
Serologic Outcomes | Outcome measure will be assessed at 6, 12 , and up to 18 months after enrollment.
  HIV antibody testing is performed at the baseline and semi-annual follow-up visits using standard ELISA screening and confirmatory Western Blots. In addition, Hepatitis B and C antibody testing is performed at baseline and follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: William W. Latimer, PhD, MPH, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Baltimore, Maryland, United States